CLINICAL TRIAL: NCT01393600
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled, Two-Period Cross-Over Study to Evaluate the Efficacy and Safety of NBI-98854 for the Treatment of Tardive Dyskinesia in Subjects With Schizophrenia or Schizoaffective Disorder
Brief Title: NBI-98854 for the Treatment of Tardive Dyskinesia in Subjects With Schizophrenia or Schizoaffective Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NBI-98854-1101
Record Dates: First submitted 2011-07-11; First posted 2011-07-13 (Estimated); Results first posted 2017-08-10 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-07

CONDITIONS: Tardive Dyskinesia
MeSH Terms: conditions — Tardive Dyskinesia | interventions — valbenazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NBI-98854 12.5 mg (Experimental): During the Cross-Over Study, subjects will be randomly assigned to receive one of the following treatment sequences:
  Sequence 1: Placebo once daily dose for Days 1-14 and 12.5 mg NBI-98854 once daily dose for Days 15-28.
  Sequence 2: 12.5 mg NBI-98854 once daily dose for Days 1-14 and placebo once daily dose for Days 15-28.
  Interventions: Drug: NBI-98854; Drug: Placebo
- NBI-98854 50 mg (Experimental): During the Cross-Over Study, subjects will be randomly assigned to receive one of the following treatment sequences:
  Sequence 3: Placebo once daily dose for Days 1-14 and 50 mg NBI-98854 once daily dose for Days 15-28.
  Sequence 4: 50 mg NBI-98854 once daily dose for Days 1-14 and placebo once daily dose for Days 15-28.
  Interventions: Drug: NBI-98854; Drug: Placebo

INTERVENTIONS:
Drug: NBI-98854 — 12.5 mg powder in bottle once daily for 14 days
  Arms: NBI-98854 12.5 mg
Drug: NBI-98854 — 50 mg powder in bottle once daily for 14 days
  Arms: NBI-98854 50 mg
Drug: Placebo — Solution containing no active substance

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of two doses (12.5 and 50 mg) of NBI-98854 administered once daily (q.d.) for the treatment of tardive dyskinesia in subjects with schizophrenia or schizoaffective disorder.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of schizophrenia or schizoaffective disorder and a clinical diagnosis of neuroleptic-induced tardive dyskinesia as defined in the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV), 333.82 (see Appendix 17.1) for at least 3 months prior to screening.
* Be receiving a stable dose of antipsychotic medication for a minimum of 30 days before study start. Subjects who are not using antipsychotic medication must have stable psychiatric status.
* Have the doses of concurrent medications and the conditions being treated be stable for a minimum of 30 days before study start and be expected to remain stable during the study.
* Subjects of childbearing potential must agree to use hormonal or two forms of nonhormonal birth control during the study.
* Female subjects must not be pregnant.
* Be in good general health and expected to complete the clinical study as designed.
* Have a body mass index (BMI) of 18 to 38 kg/m2 (both inclusive).
* Have adequate hearing, vision, and language skills to perform the procedures specified in the protocol.
* Have a negative urine drug screen (negative for amphetamines, barbiturates, benzodiazepine, phencyclidine, cocaine, opiates, or cannabinoids) at screening and study start, except for any subject receiving a stable dose of benzodiazepine.
* Have a negative alcohol breath test at screening and study start.

Exclusion Criteria:

* Have an active clinically significant unstable medical condition within 1 month (30 days) prior to screening.
* Have a history of substance dependence or substance (drug) or alcohol abuse within the 3 months before study start(nicotine and caffeine dependence are not exclusionary).
* Have a known history of neuroleptic malignant syndrome.
* Have a significant risk of suicidal or violent behavior.
* Receiving any excluded concomitant medication such as reserpine, metoclopramide, stimulants, or tetrabenazine
* Receiving medication for the treatment of tardive dyskinesia.
* Have a positive human immunodeficiency virus antibody, (HIV-Ab), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody result at screening or have a history of positive result.
* Have received an investigational drug within 30 days before screening or plan to use an investigational drug (other than NBI-98854) during the study.
* Have an allergy, hypersensitivity, or intolerance to tetrabenazine.
* Have had previous exposure with NBI-98854.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher O'Brien, MD, Study Director — Neurocrine Biosciences
Locations (11):
- United States (11):
  - Woodland International Research Group, Inc, Little Rock, Arkansas
  - Synergy Clinical Research, National City, California
  - UCSD Outpatient Psychiatry, San Diego, California
  - PCSD - Feighner Research, San Diego, California
  - San Marcus Research Clinic, Inc., Miami, Florida
  - Medical Research Marseilles, Miami, Florida
  - Scientific Clinical Research, Inc., North Miami, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - St. Louis Clinical Trials, St Louis, Missouri
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - CAMC Clinical Trials Center, Charleston, West Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients with a clinical diagnosis of schizophrenia or schizoaffective disorder with moderate or severe symptoms of tardive dyskinesia (TD) from 10 centers in the United States. The last patient completed in February 2012.
Groups:
- Placebo, Then Valbenazine 12.5 mg: Participants first received Placebo (matching valbenazine solution) once daily from Day 1 to 14, then they received valbenazine 12.5 mg solution once daily from Day 15 to 28.
- Valbenazine 12.5 mg, Then Placebo: Participants first received valbenazine 12.5 mg solution once daily from Day 1 to 14, then they received Placebo (matching valbenazine solution) once daily from Day 15 to 28.
- Placebo, Then Valbenazine 50 mg: Participants first received Placebo (matching valbenazine solution) once daily from Day 1 to 14, then they received valbenazine 50 mg solution once daily from Day 15 to 28.
- Valbenazine 50 mg, Then Placebo: Participants first received valbenazine 50 mg solution once daily from Day 1 to 14, then they received Placebo (matching valbenazine solution) once daily from Day 15 to 28.
Period: Treatment Period 1 (Day 1 to 14)
Arm/Group | Placebo, Then Valbenazine 12.5 mg | Valbenazine 12.5 mg, Then Placebo | Placebo, Then Valbenazine 50 mg | Valbenazine 50 mg, Then Placebo
Started | 9 | 8 | 10 | 10
Completed | 9 | 7 | 9 | 9
Not Completed | 0 | 1 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1
Period: Treatment Period 2 (Day 15 to 28)
Arm/Group | Placebo, Then Valbenazine 12.5 mg | Valbenazine 12.5 mg, Then Placebo | Placebo, Then Valbenazine 50 mg | Valbenazine 50 mg, Then Placebo
Started | 9 | 7 | 9 | 9
Completed | 9 | 7 | 7 | 8
Not Completed | 0 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Period: Follow-up Period (Day 29 to 35)
Arm/Group | Placebo, Then Valbenazine 12.5 mg | Valbenazine 12.5 mg, Then Placebo | Placebo, Then Valbenazine 50 mg | Valbenazine 50 mg, Then Placebo
Started | 9 | 7 | 7 | 8
Completed | 9 | 7 | 6 | 8
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: All randomized subjects who received at least one dose of study drug.
Arm/Group | All Subjects
Number analyzed (Participants) | 37
Age, Continuous [Mean (Full Range); unit: years] | 51.1 [29 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 12
  Caucasian | 15
  Hispanic | 10
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 29.9 [18.1 to 42.0]
Age of Schizophrenia/Schizoaffective Disorder Diagnosis [Mean (Full Range); unit: years] | 25.8 [8 to 54]
Age at TD Diagnosis [Mean (Full Range); unit: years] | 41.7 [18 to 63]

OUTCOME MEASURES:

1. Primary Outcome: Abnormal Involuntary Movement Scale (AIMS) Dyskinesia Total Score
Description: Severity of TD symptoms assessed by AIMS dyskinesia total score (sum of items 1 through 7), as assessed by blinded central AIMS video raters. The AIMS Total Dyskinesia Score rates a total of 7 items, rating involuntary movement from 0 (no dyskinesia) to 4 (severe dyskinesia). Items 1 through 7 include facial and oral movements (Items 1-4), extremity movements (Items 5-6), and trunk movements (Item 7). The AIMS dyskinesia total score for Items 1-7 ranges from 0 to 28; a higher score reflects increased severity.
Time Frame: Day 15 and 29, averaged
Population: Intent to treat (ITT) analysis set (all subjects who received at least 8 doses of study drug during Treatment Period 1 and had an AIMS dyskinesia total score value for Day 15).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Placebo (matching valbenazine solution)
- Valbenazine 12.5 mg: Valbenazine 12.5 mg solution
- Valbenazine 50 mg: Valbenazine 50 mg solution
Arm/Group | Placebo | Valbenazine 12.5 mg | Valbenazine 50 mg
Number analyzed (Participants) | 33 | 17 | 15
units on a scale | 9.9 (0.7) | 9.1 (1.2) | 8.8 (1.2)
Statistical Analysis 1: Comparison: Placebo vs Valbenazine 12.5 mg; Test type: Other; p = 0.5880, ANOVA; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-3.3 to 1.9], Standard Error of Mean 1.3
Statistical Analysis 2: Comparison: Placebo vs Valbenazine 50 mg; Test type: Other; p = 0.4184, ANOVA; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-3.8 to 1.6], Standard Error of Mean 1.3

2. Secondary Outcome: Clinical Global Impression - Global Improvement of TD (CGI-TD)
Description: Clinician's perspective of the participant's overall improvement of TD symptoms over time. The CGI-TD is based on a 7-point scale (range: 1=very much improved to 7=very much worse).
Time Frame: Day 15 and 29, averaged
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Valbenazine 12.5mg Placebo: Participants who received Placebo (matching valbenazine 12.5mg solution) once daily from Day 1 to 14 and participants who received Placebo (matching valbenazine 12.5mg solution) from Day 15 to 28.
- Valbenazine 12.5mg: Participants who received valbenazine 12.5mg solution once daily from Day 1 to 14 and participants who received valbenazine 12.5mg solution from Day 15 to 28.
- Valbenazine 50mg Placebo: Participants who received Placebo (matching valbenazine 50mg solution) once daily from Day 1 to 14 and participants who received Placebo (matching valbenazine 50mg solution) from Day 15 to 28.
- Valbenazine 50mg: Participants who received valbenazine 50mg solution once daily from Day 1 to 14 and participants who received valbenazine 50mg solution from Day 15 to 28.
Arm/Group | Valbenazine 12.5mg Placebo | Valbenazine 12.5mg | Valbenazine 50mg Placebo | Valbenazine 50mg
Number analyzed (Participants) | 16 | 17 | 17 | 15
units on a scale | 2.2 (0.2) | 2.2 (0.2) | 3.2 (0.3) | 2.6 (0.3)

3. Post Hoc Outcome: Abnormal Involuntary Movement Scale (AIMS) Dyskinesia Total Score for Combined NBI-98854 Dose Groups (Excluding 1 Site)
Description: as for outcome 1
Time Frame: Day 15 and 29, averaged
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Valbenazine 12.5 mg | Valbenazine 50 mg
Number analyzed (Participants) | 26 | 15 | 10
units on a scale | 10.3 (0.9) | 9.9 (1.1) | 6.1 (1.2)
Statistical Analysis 1: Comparison: Placebo vs Valbenazine 12.5 mg; Test type: Other; p = 0.6761, ANOVA; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-2.4 to 1.6], Standard Error of Mean 1.0
Statistical Analysis 2: Comparison: Placebo vs Valbenazine 50 mg; Test type: Other; p = 0.0015, ANOVA; Mean Difference (Final Values) = -4.2, 95% CI 2-sided [-6.6 to -1.8], Standard Error of Mean 1.1

ADVERSE EVENTS:
Time Frame: up to 35 days
Groups:
- Placebo: Placebo (matching NBI-98854 solution) for 28 days followed by 7 days of posttreatment.
- NBI-98854 12.5 mg: NBI-98854 12.5 mg solution for 28 days followed by 7 days of posttreatment.
- NBI-98854 50 mg: NBI-98854 50 mg solution for 28 days followed by 7 days of posttreatment.
Arm/Group | Placebo | NBI-98854 12.5 mg | NBI-98854 50 mg
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/17 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/35 | 1/17 | 0/19
Other Adverse Events (participants affected / at risk) | 4/35 | 4/17 | 6/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=35) | NBI-98854 12.5 mg (N=17) | NBI-98854 50 mg (N=19)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=35) | NBI-98854 12.5 mg (N=17) | NBI-98854 50 mg (N=19)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (4) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Urine analysis abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Akathisia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (5) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sedation (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the PI has the right to publish results provided such publication does not violate confidentiality or IP provisions within the contract with the Sponsor. Prior to submission for publication or presentation of results, the PI must provide the Sponsor time for review. The Sponsor can request the PI to withhold or remove information from all publications. For a multi-center study, any publication of results by the PI shall not be made before the first multi-center publication.